CLINICAL TRIAL: NCT03738540
Title: Pilot Randomized Trial of a Telephone Weight Loss, Nutrition, Exercise Study (WeLNES)
Brief Title: Pilot Trial of a Telephone Weight Loss, Nutrition, Exercise Study
Acronym: WeLNES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 8693; NCI-2019-02521 (Registry Identifier: NCI / CTRP); RG1001915 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-10-02; First posted 2018-11-13 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Weight Loss; Weight, Body
Keywords: Weight loss; Nutrition; Exercise; Diet; Telephone coaching
MeSH Terms: conditions — Weight Loss; Body Weight; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): This is the experimental arm of the study. This includes 25 weekly then biweekly sessions of experimental therapy via telephone. Therapy description withheld to protect the integrity of the study.
  Interventions: Behavioral: TALK study group
- Control (Active Comparator): This is the control arm of the study. This includes This includes 25 weekly then biweekly sessions of control therapy via telephone.Therapy description withheld to protect the integrity of the study.
  Interventions: Behavioral: TALK control group

INTERVENTIONS:
Behavioral: TALK study group — Telephone Delivered Intervention
  Arms: Experimental
Behavioral: TALK control group — Telephone Delivered Intervention
  Arms: Control

SUMMARY:
Many behavioral weight loss interventions have been developed, but still have significant limitations in terms of achieving clinically significant, sustained weight loss. A recent study incorporating Acceptance and Commitment Therapy (ACT) in a randomized clinical trial resulted in participants who attained significantly greater 12-month weight loss in the ACT arm than those assigned to standard behavioral treatment, suggesting that ACT may have the potential to improve behavioral weight loss outcomes. The investigators have developed a novel telephone-delivered version of the ACT behavioral weight loss intervention, based on proven success using ACT telephone counseling intervention for smoking cessation.

DETAILED DESCRIPTION:
There is consistent evidence from observational studies that higher amounts of body fat are associated with increased risks of cancer. Many behavioral weight loss interventions have been developed, but still have significant limitations in terms of achieving clinically significant, sustained weight loss. A recent study incorporating Acceptance and Commitment Therapy (ACT) in a randomized clinical trial resulted in participants who attained significantly greater 12-month weight loss in the ACT arm than those assigned to standard behavioral treatment, suggesting that ACT may have the potential to improve behavioral weight loss outcomes. However, this study required in-person clinic visits with treatment groups, which limits its potential reach and disseminability. The investigators have developed a novel telephone-delivered version of the ACT behavioral weight loss intervention, based on our proven success using ACT telephone counseling intervention for smoking cessation. There will be a two-arm pilot randomized trial (N = 100), comparing the ACT telephone intervention to a standard behavioral treatment (SBT) telephone control. The pilot RCT will yield engagement, receptivity, and preliminary weight loss results that will provide critical and timely weight loss intervention data.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older,
* overweight or obese (BMI ≥ 27),
* wants to lose weight through healthy behavior change, beginning in the next 30 days,
* interested in learning skills to lose weight,
* willing to be randomly assigned to either condition,
* resides in US,
* has daily access to their own phone and email,
* does not have a medical or psychiatric condition that would limit their ability to comply with the behavioral recommendations of the program or pose a risk to the participant during weight loss, including meeting criteria for binge eating disorder,
* not pregnant or planning to become pregnant in the next 12 months,
* in the past 3 months changed the dosage of prescription medications that can cause a significant change in weight or appetite,
* have lost more than 5% of their weight in the past 6 months,
* willing and able to read in English,
* not participating in or planning to participate in other weight loss programs, and
* has not participated in our other ACT interventions. To increase follow-up data retention, eligibility criteria also include:
* willing to complete the follow-up survey, and (16) provide email, phone, and mailing address.

Exclusion Criteria:

* Opposite of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
12-month weight loss | 12 months post randomization
  Weight loss measured by BodyTrace scale. The BodyTrace medical body weight scale is a physical scale capable of assessing weight from 0.2 lbs to 397 lbs (0.1 kg to 180 kg) and securely sending data remotely through cellular (GSM) network.

SECONDARY OUTCOMES:
3-month weight loss | 3 months post randomization
  Weight loss measured by BodyTrace scale. The BodyTrace medical body weight scale is a physical scale capable of assessing weight from 0.2 lbs to 397 lbs (0.1 kg to 180 kg) and securely sending data remotely through cellular (GSM) network.
6-month weight loss | 6 months post randomization
  Weight loss measured by BodyTrace scale. The BodyTrace medical body weight scale is a physical scale capable of assessing weight from 0.2 lbs to 397 lbs (0.1 kg to 180 kg) and securely sending data remotely through cellular (GSM) network.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Bricker, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bricker JB, Mull KE, Sullivan BM, Forman EM. Efficacy of telehealth acceptance and commitment therapy for weight loss: a pilot randomized clinical trial. Transl Behav Med. 2021 Aug 13;11(8):1527-1536. doi: 10.1093/tbm/ibab012. PMID 33787926
- See also: Study recruitment website — http://welnes.org